CLINICAL TRIAL: NCT06091072
Title: Feasibility of in Vivo Image-guided Navigation During Robotic Sentinel Node Removal
Brief Title: Image-guided Navigation During Robotic Sentinel Node Removal
Acronym: N21LND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL77462.031.21
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Intervention Model Description: One group to evaluate the feasibility of the proposed method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients scheduled for sentinel node procedure (Experimental): This is a single-center observational feasibility study to evaluate the overall performance of the surgical navigation system during robotic surgery, without impact on the surgical procedure itself. The duration of this study will be approximately 2.5 years. Patients scheduled for a sentinel node procedure at the NKI are eligible for inclusion. Patients are informed about the study before the planned surgery and, after being provided with the necessary information regarding participation in the study, will be asked for informed consent. No additional risk is expected using the NDI navigation setup. Patients will receive some additional radiation due to the CT scan during surgery; a perioperative CBCT scan (~ 4 mSv) is acquired. This extra dose is low, considering other standard imaging in these patients like, pre-operative imaging with SPECT/CT scans. After surgery, no further participation or cooperation of the patient is required.
  Interventions: Other: Image-guided navigation

INTERVENTIONS:
Other: Image-guided navigation — A patient-specific 3D model will be created using an available pre-operative SPECT/CT scan. Pre-operatively, three electromagnetic patient trackers will be attached to the patients' skin, close to the pelvis, allowing tracking the patient's position during surgery. After anesthesia and before the skin disinfection procedure, the patient is placed in the final surgical position, where an intra-operative CBCT scan is performed required for the image-guided surgery workflow. During surgery, the preoperative images and 3D model will be visible for the surgeon together with a blunt-tip electromagnetic pointer enabling surgical navigation during robotic surgery. Anatomical structures will be used to validate the accuracy of the navigation. When the target is identified by the surgeon, the pointer is used to store the location digitally. Scheduled standard clinical 99mTc will be used as validation for target(s) identification.

SUMMARY:
Image-guided navigation based on pre-operative imaging can give the surgeon more insight into the location of the sentinel nodes in relation to other anatomical structures. The purpose of the study is to investigate the feasibility of image-guided navigation during robot-assisted surgery to treat cancer in the pelvic area.Ultimately, the application of navigation during robot-assisted sentinel node dissection could potentially improve the outcome of surgery for the patient.

DETAILED DESCRIPTION:
Image-guided navigation surgery allows for full utilization of pre-operative imaging during surgery, and has the potential of reducing both irradical resections and morbidity. It has successfully been applied in the AvL for open abdominal surgery, however more and more surgeries are being performed less invasive using robot surgery. Rapid extension of robot-assisted surgery has increased the need for robot-compliant image-guided techniques.

Unfortunately, tactile feedback is lacking in these robotic surgeries, which increases the additional value of image-guided navigation. In this study, patients will undergo an abdominal sentinel node dissection in order to evaluate the actual technical benefit of robotic navigation. This is the first feasibility study towards clinical implementation of the navigation setup into robot-assisted image-guided navigation surgery. The results of this study will be the base for new studies, evaluating the clinical benefit of image-guided navigation for robot surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for abdominal robotic sentinel node resection
* ≥ 18 years old
* Provided written 'informed consent'
* Sentinel nodes should be fixed relative to retroperitoneal structures or major vessels.

Exclusion Criteria:

* Metal hip implants / implants in the pelvic area
* Pacemaker, defibrillator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of image-guide assisted sentinel node removal | One day
  The percentage of successful image-guide assisted sentinel nodes removed, in which failure is defined as sentinel nodes which are per-operatively incorrectly identified as target SN by the navigation.

SECONDARY OUTCOMES:
Usability of image-guided navigation | One day
  Evaluation of the usability of the image-guided navigation will be evaluated using the system usability scale (SUS). This scale ranges from 0-100 where a higher score means a better outcome.
Time | One day
  Time to localization and removal of the sentinel node and total surgical time will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No